CLINICAL TRIAL: NCT01106144
Title: Genetic Predictive Model Based on Single Nucleotide Polymorphisms in the DNA Repair Pathway and Drug Metabolis/Transport Pharmacogenetics in the Prediction of Response and Treatment Outcomes in Acute Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan Kim, Division of Hematology and Oncology/Samsung Medical Center/Sungkyunkwan University
Other Study IDs: 2008-08-094
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Patients With Acute Myeloid Leukemia; Patients Receiving Induction/Consolidation Chemotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Preserved bone marrow sample from the adult patients with acute myeloid leukemia
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute myeloid leukemia

SUMMARY:
The main component in the treatment of acute myeloid leukemia (AML) is consist of anthracycline (such as daunorubicin or idarubicin) and cytarabine. Inter-individual variability of transport/metabolism of the chemotherapeutic agent and several genetic pathways involved in the drug action might be associated with different response following the treatment for AML usually consisted of chemotherapy and/or transplantation. One of potential pathways involved in the drug action is DNA repair pathway, accordingly single nucleotide polymorphisms (SNPs) in the DNA repair machinery pathway might be a predictive marker for therapy outcomes in AML.

Several genes were involved in the DNA repair machinery which are 1) Nonhomologous end joining (NHEJ) pathway involved in the G1/S phase, 2) Homologous recombinational repair (HRR) pathway involved in the S/G2 phase. XRCC4, LIG4, MRN and ATM are well known genes involved in the NHEJ pathway, while MRE11, RAD50, NBS1 (MRN), RAD51, XRCC2, XRCC3, RAD51B, RAD51C, RAD 51D, RAD52 or RAD54 are known to be associated with HRR pathway.

A study suggested that the SNPs in the DNA repair pathway was involved in the susceptibility of secondary AML developing after chemotherapy or autologous hematopoietic stem cell transplantation, thus these SNP markers could become a predictive marker for secondary AML. However, it has never been investigated for multiple candidate pathways simultaneously with relateively larger number of patients. Accordingly, the current study attempts to investigate the potential role of the genotype markers in multiple candidate pathways, esp. focused on the DNA repair machinery, with respect to response following chemotherapy or survival of AML patients.

Total of over 500 archived samples from the patients diagnosed as acute myeloid leukemia at the Samsung Medical Center, Seoul, Korea will be included, and genomic DNAs will be extracted and will be examined for their genotypes of the candidate SNPs involved in the DNA repair pathways. Then statistical analysis will be pursued for single marker analysis, haplotype analysis and for the construction of genetic risk model based on the multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute myeloid leukemia
* 15 years or older
* patients treated with induction/consolidation chemotherapy
* patients with available bone marrow sample

Exclusion Criteria:

* acute biphenotypic leukemia

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with acute myeloid leukemia receiving induction/consolidation combination chemotherapy at Samsung Medical Center from 1996 to 2005
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-05

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center IRB, Seoul, South Korea, South Korea